CLINICAL TRIAL: NCT05926557
Title: Treatment of Peri-implant Mucositis by Non-surgical Debridement and Additional Application of a Spermidine-based Gel
Brief Title: Treatment of Peri-implant Mucositis by Application of a Spermidine-based Gel
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Luca Ramaglia, Clinical Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 249/2023
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-02

CONDITIONS: Peri-implant Mucositis; Mucositis Oral
Keywords: Peri-implant Mucositis; Spermidine
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Intervention Model Description: The study will be designed as a double-arm randomized controlled clinical trial. Mucositis will be treated with spermidine gel + non-surgical debridement (NSMD) in Test group and with NSMD alone in Control group. All clinical parameters will be recorded at baseline, 1 and 3 months.
Who Masked: Investigator, Outcomes Assessor
Masking Description: All patients are not masked with respect to test and control procedures, with prior written informed consent. So, they will be divided in the two groups of study after a process of randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spermidine Group (Experimental): Mechanical therapy (NSMD) will be performed by means of an ultrasonic scaler with a plastic tip. Finally, the spermidine-based gel will be applied in the peri-implant sulcus using a blunt-tipped needle.
  Interventions: Procedure: Spermidine gel
- NSMD Group (Active Comparator): Control group will be treated only through a non-surgical mechanical therapy with curettes or scaler peek tips.
  Interventions: Procedure: NSMD

INTERVENTIONS:
Procedure: Spermidine gel — First step: Non-surgical mechanical debridement (NSMD) Second step: application of spermidine gel
  Arms: Spermidine Group
Procedure: NSMD — Only mechanical debridement with curettes and scaler peek tips
  Arms: NSMD Group

SUMMARY:
The aim of the study is to evaluate the potential of a spermidine-based topical gel as an adjuvant to non-surgical treatment of peri-implant mucositis. After a meticulous selection, patients will be randomly assigned to Test (spermidine gel + non-surgical debridement) or Control group (non-surgical debridement).

DETAILED DESCRIPTION:
Following the recording of the clinical parameters (BoP, FMPS, FMBS, PD), mechanical therapy (NSMD) will be performed in the Test group (spermidine gel) by means of an ultrasonic scaler with a plastic tip. Finally, the spermidine-based gel will be applied in the peri-implant sulcus using a blunt-tipped needle. Control group will instead be treated only through the NSMD.

Finally, after 3 months the clinical parameters (BoP, FMPS, FMBS, PD) will be recorded again and the final evaluation will be performed. Data analysis will be performed using statistical software.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Non-smokers and smokers ( ≤ 10 cigarettes/day);
* Presence of at least 1 implant in mucositis, clinically and radiographically detected;
* The implant in mucositis (tissue-level or bone-level) must support a fixed prosthetic device (single crown), cemented or screwed.

Exclusion Criteria:

* Cancer patients;
* Periodontally Compromised Patients;
* Uncontrolled diabetic patients;
* Prolonged antibiotic treatment or anti-inflammatory treatment in the previous 6 months;
* Pregnant or breastfeeding patients;
* Implants that support mobile prosthetic products;
* Implants in peri-implantitis, detected clinically and radiographically.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change of BoP (+/-) | baseline, 1 and 3 months after periodontal therapy
  Bleeding on periodontal probing

SECONDARY OUTCOMES:
Change of Full-mouth Plaque Score (FMPS; %) | baseline, 1 and 3 months after periodontal therapy
  Percentage of all sites exhibiting plaque
Change of Full-mouth Bleeding Score (FMBS; %) | baseline, 1 and 3 months after periodontal therapy
  Percentage of all sites exhibiting bleeding
Change of Probing Depth (PD; millimeters) | baseline, 1 and 3 months after periodontal therapy
  Distance from the gingival margin to the bottom of the peri-implant pocket

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: No